CLINICAL TRIAL: NCT01693536
Title: Effective Change of Behaviour of the Elderly in Normal General Practice
Brief Title: Can Primary Care Change Elderly Physical Activity and Salt Intake? An Australian Pilot Trial
Acronym: ECOBEING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health HQ (Other)
Responsible Party: Principal Investigator, Norman Hohl, Medical Director, Health HQ
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RO783
Record Dates: First submitted 2012-09-16; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Health Behaviour
Keywords: Elderly; Sodium reduction; Fitness increase; Primary Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counselling (Experimental): Three dietician visits focussed on education to find food with sodium less than 120mg/100gms.
  Two physiotherapist visits focussed on teaching personalised sustainable practical exercise.
  Interventions: Behavioral: Lifestyle counselling
- Control (No Intervention): Control group was offered free skin cancer check and wait listed for the same lifestyle counselling after the six months of the study.

INTERVENTIONS:
Behavioral: Lifestyle counselling — as in Arm Description
  Other Names: salt reduction in the elderly; increased fitness in the elderly
  Arms: Lifestyle counselling

SUMMARY:
A randomised controlled trial to test if offering three visits to a dietician + two visits to a physiotherapist over six months + a home sphygmomanometer, will result in a reduction in sodium intake and an increase in fitness in people over 75yrs. Volunteers were enrolled from Oct 2008 to July 2009.

DETAILED DESCRIPTION:
There is evidence that both sedentary lifestyle and high sodium diets contribute to cardiovascular disease and possibly dementia among the elderly. There is a need to show that minimal intervention can reduce sodium intake and increase fitness in the elderly. Finland has shown that five dietician visits/year could change diet in respect to fat and fibre. In Australia the National Health Insurer (Medicare) funds five allied health visits/year for those with chronic disease, hence our use of this model. This is consistent with WHO guidelines for a national approach using existing health infrastructure. The elderly (75-95yrs) were chosen as this group is thought most difficult to change behaviour and has a higher incidence of dementia.

ELIGIBILITY:
Inclusion Criteria:

* Living independently
* Must be able to walk for six minutes

Exclusion Criteria:

* Dementia as defined by Standardised Mini-Mental State Examination score <25/30
* All patients of HealthHQ-Southport General Practice

Ages: 75 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
the change in morning urine sodium/potassium ratio | between enrollment and six months
  this measure is to reflect sodium intake. A 24hr urinary sodium cannot be readily validated as an accurate collection and even in the Trials of Hypertension Prevention study was changed to 8hrs to assist compliance. A spot morning ratio is a useful marker of sodium intake for group evaluation.
the increased distance in a six minute walk test | between enrollment and six months
  to measure objectively an increase in fitness the increase in the six minute walk test was used

SECONDARY OUTCOMES:
change in systolic BP | between enrollment and six months
  teaching people to reduce sodium intake and increase fitness may reduce systolic blood pressure as a secondary outcome
change in doses/day of antihypertensive medication | between enrollment and six months
  teaching reduction in sodium and increased fitness may mean people need less antihypertensive medication as a secondary outcome
change in waist measurement | between enrollment and six months
  teaching increased fitness would be expected to reduce waist measurement as a secondary outcome
change in weight & BMI | between enrollment and six months
  teaching increased fitness would be expected to reduce weight and therefore calculated Body Mass Index as a secondary outcome
change in cognition measurement | between enrollment and six months
  Cognition measurements using the Standardised Mini-Mental State Examination, and the more comprehensive and sensitive Addenbrooke Cognitive Examination to compare those in the intervention group with the highest and lowest quartiles of reduction in sodium intake + increased fitness (equally weighted), as a secondary outcome of teaching these lifestyle changes.

CONTACTS AND LOCATIONS:
Overall Officials: Norman A Hohl, MBBS, FRACGP, Principal Investigator — Medical Director Health HQ, Ass Prof Bond Uni Faculty Health Science; Chris del Mar, FAFPHM,MD,MA, Study Chair — Dean BOND Uni Faculty Health Science & Medicine (at time of study)
Locations (1):
- Health HQ-Southport General Practice, Southport, Queensland, Australia

REFERENCES:
- [Background] Cook NR, Cutler JA, Obarzanek E, Buring JE, Rexrode KM, Kumanyika SK, Appel LJ, Whelton PK. Long term effects of dietary sodium reduction on cardiovascular disease outcomes: observational follow-up of the trials of hypertension prevention (TOHP). BMJ. 2007 Apr 28;334(7599):885-8. doi: 10.1136/bmj.39147.604896.55. Epub 2007 Apr 20. PMID 17449506
- [Background] Lindstrom J, Ilanne-Parikka P, Peltonen M, Aunola S, Eriksson JG, Hemio K, Hamalainen H, Harkonen P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Mannelin M, Paturi M, Sundvall J, Valle TT, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. Sustained reduction in the incidence of type 2 diabetes by lifestyle intervention: follow-up of the Finnish Diabetes Prevention Study. Lancet. 2006 Nov 11;368(9548):1673-9. doi: 10.1016/S0140-6736(06)69701-8. PMID 17098085
- [Background] Joint Health Surveys Unit (NatCen and UCL). A survey of 24 hour and spot urinary sodium and potassium excretion in a representative sample of the Scottish population. Food Standards Agency Scotland, 2007